CLINICAL TRIAL: NCT04258280
Title: Parent Communication Study IV: Improving Genetic Counseling for BRCA+ Mothers
Brief Title: Improving Genetic Counseling for BRCA+ Mothers
Acronym: PCS IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 00001137
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator)
  Interventions: Behavioral: Education
- Enhanced Care (Experimental)
  Interventions: Behavioral: Education and counseling

INTERVENTIONS:
Behavioral: Education and counseling — Education includes a workbook, counseling includes peer support.
  Arms: Enhanced Care
Behavioral: Education — Education includes a workbook.
  Arms: Usual Care

SUMMARY:
Genetic counseling and testing for hereditary breast cancer may reveal that you, and possibly your blood relatives, are at increased risk for the disease across the lifespan. This includes biological children, both male and female. We do not yet know the best ways to educate mothers who have a risk gene (are BRCA+) about whether, when, and how to share genetic information with their children or manage their thoughts and feelings. The purpose of this study is to help mothers make more informed choices about talking with children about hereditary breast cancer, provide them with age-and gender-appropriate information and emotional support, and improve their psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Mothers/primary caregivers to adolescents/young adults ages 13-24 years-old.
* Participating in genetic testing for hereditary breast cancer.
* Adequately speak/read English.

Exclusion Criteria:

- Does not meet inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Communication | 1- and 6-months post-treatment
  Parent-child and family communication of hereditary cancer risk.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States